CLINICAL TRIAL: NCT02511743
Title: Knowledge and Practice of Chinese Medical Specialists Regarding Chronic Hepatitis B Virus
Brief Title: Knowledge and Practice of Chinese Medical Specialists Regarding Chronic Hepatitis B Virus Infection
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Guiqiang Wang, Professor in Medicine, Peking University First Hospital
Other Study IDs: 2015[888]
Record Dates: First submitted 2015-05-04; First posted 2015-07-30 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Physicians

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- physicians: physicians taking care of patients with chronic Hepatitis B Virus infection
  Interventions: Other: physicians

INTERVENTIONS:
Other: physicians — physicians taking care of patients with chronic Hepatitis B Virus infection, without intervention

SUMMARY:
The aim of this study was to evaluate knowledge and behavior of physicians regarding Hepatitis B Virus. The investigators designed a 30-item self-administered questionnaire assessing physicians' knowledge and behavior regarding chronic Hepatitis B Virus infection. These results provide data support for updating guidelines, continuing training, and even developing policies in medical insurance.

DETAILED DESCRIPTION:
Schedule of the study:

Before March 1, 2015: study design, completing questionnaire design, and all preparatory work; Before July 1, 2015: a kick-off meeting for plot study, modifying the questionnaire, and obtaining all the questionnaires; Before September 30, 2015: finishing data entry, statistical analysis, drafting the report, and issued a final report

ELIGIBILITY:
Inclusion Criteria:

1. Mainly engaged in liver disease diagnosis and treatment;
2. Diagnosis and treatment at least 10 patients with chronic Hepatitis B Virus infection per week.

Exclusion Criteria:

1. young doctors working in less than one year;
2. physicians working in hospital of Traditional Chinese Medicine
3. visiting doctors.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: physicians fullfill the following criterion:
  1. Mainly engaged in liver disease diagnosis and treatment;
  2. Diagnosis and treatment at least 10 patients with chronic Hepatitis B Virus infection per week.
Sampling Method: Non-Probability Sample
Enrollment: 2871 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
30-item self-administered questionnaire assessing physicians' knowledge and behavior regarding chronic Hepatitis B Virus infection. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: guiqiang wang, M.D., Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China